CLINICAL TRIAL: NCT04220476
Title: CIMER: Combined Immunotherapies in Metastatic ER+ Breast Cancer
Acronym: CIMER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Initiating a new study with revised Statistics.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-09020752
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: metastatic Breast cancer; HR+HER2-; HR + BC; SBRT
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARM 1 - Letrozole and Palbociclib (Active Comparator): Patients randomized to arm 1 will start standard Letrozole followed by Palbociclib at day 21.
  Interventions: Drug: Letrozole 2.5Mg Tab; Drug: Palbociclib 125mg
- ARM 2 - Letrozole and Palbociclib + I-SBRT (Active Comparator): Patients randomized to arm 2 will start letrozole alone, and add palbociclib on day 21, after completion of I-SBRT. Treatment may be given daily (to keep the total I-SBRT treatment time to ≤ 12 days) and lesions targeted with I-SBRT will thus be alternated each day to accommodate for the 48 hour interval between fractions.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT) (50GY in 5 fractions); Drug: Letrozole 2.5Mg Tab; Drug: Palbociclib 125mg

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) (50GY in 5 fractions) — Patients randomized to arm 2 will start letrozole alone, and add palbociclib on day 21, after completion of I-SBRT. They will undergo tumor Immunogenic-SBRT(I-SBRT) days 1-12 (+/-2 days, to enable inclusion of holidays). During the week preceding day 1, they will undergo simulation and planning for radiotherapy. Each oligometastatic lesion will be treated with I-SBRT every 48 hours. Treatment may be given daily (to keep the total I-SBRT treatment time to ≤ 12 days) and lesions targeted with I-SBRT will thus be alternated each day to accommodate for the 48 hour interval between fractions
  Arms: ARM 2 - Letrozole and Palbociclib + I-SBRT
Drug: Letrozole 2.5Mg Tab — All patients start standard therapy with oral letrozole (Femara), day 1 of the study.
Drug: Palbociclib 125mg — Patients randomized to arm 2 will start letrozole alone, and add palbociclib on day 21, after completion of I-SBRT.

SUMMARY:
Women with Hormone Receptor (HR)+ Human Epidermal growth factor Receptor (HER)2- metastatic breast cancer are eligible to a randomized trial. Patients receiving standard first line therapy for metastatic HR+ Breast cancer(BC) (letrozole+palbociclib) are randomly assigned to also receive Stereotactic Body Radiation Therapy(SBRT) to each metastatic lesion.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years of age pre and post-menopausal
* Oligometastatic disease (≤ 5 sites of disease)
* Premenopausal status is defined as either:
* Patient had last menstrual period within the last 12 months, OR
* If on tamoxifen or toremifene within the past 14 days, plasma estradiol and FSH must be in the premenopausal range per local normal range, OR
* In case of therapy induced amenorrhea, plasma estradiol and/or FSH must be in the premenopausal range per local normal range.
* Patients who have undergone bilateral oophorectomy are eligible.
* Post-menopausal status defined as either 1) at least 2 years without menstrual period or 2) patients older than 50 with serological evidence of post-menopausal status or 3) hysterectomized patients of any age with FSH confirmation of post-menopausal status.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Biopsy proven diagnosis of HR+HER2- metastatic breast cancer. ER expression is >10%
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document
* Hematological WBC ≥ 2000/uL
* Absolute neutrophil count (ANC) ≥1500/µL
* Platelets ≥100 000/µL
* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Renal Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN

* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN
* Coagulation International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy if PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Active connective tissue disorders, such as lupus or scleroderma requiring flare therapy
* Current use of systemic chemotherapy, endocrine therapy or HER2-neu targeted therapy
* Male breast cancer patients
* Any lesion >5 cm in greatest diameter.
* Inability to obtain histologic proof of metastatic breast cancer
* Has received previous endocrine or chemotherapy for metastatic breast cancer.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy (second primary) that is progressing or has required active treatment within the past 3 years. Note: - - - Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patients with uncontrolled brain metastases

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Objective response rate (ORR) will be assessed. | End of study, up to 36 months.
  ORR is defined as the percentage of subjects with either a confirmed complete response (CR) or partial response (PR).
Number of Subjects achieving Progression free survival (PFS) | End of study, up to 36 months.
  Progression free survival (PFS) is defined as the time from the start of study treatment until the disease progression or death.
Number of subjects achieving Overall survival(OS) will be assessed. | End of study, up to 36 months.
  OS is defined as the time from the start of treatment until death.

SECONDARY OUTCOMES:
Serial levels of Circulating tumor DNA (ctDNA) | End of study, up to 36 months.
  serial levels ctDNA can be an early indication of progression
Circulating tumor DNA (ctDNA) levels | End of study, up to 36 months.
  Circulating tumor DNA (ctDNA) levels will be measured to determine baseline cancer heterogeneity and its response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No